CLINICAL TRIAL: NCT01920503
Title: International Registry on Cholangiocarcinoma Treatment
Acronym: CHOLANGIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Group of Endovascular Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: CHOLANGIO01; CHOLANGIO100513 (Other: IGEVO)
Record Dates: First submitted 2013-08-07; First posted 2013-08-12 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Cholangiocarcinoma
Keywords: cholangiocarcinoma; transarterial chemoembolization; doxorubicin; tumor response
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- doxorubicin: Day +1:
  Lobar Infusion ( lobe with dominant disease) of Doxorubicin preloaded into 2 ml of 70-150 µm M1 microspheres.
  Second lobar infusion of Doxorubicin preloaded into 2 ml of 70-150 µm M1 microspheres can be administered at the same time contralaterally or in a further TACE Day +30: The above procedure is repeated. Day +90: In case of response, a third administration following the above procedures will be repeated
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicina is loaded at the concentration of 50-75 mg/mq onto 2 ml of 70-150 µm M1 microspheres and is infused by TACE method
  Other Names: Adriamycin

SUMMARY:
Cholangiocarcinoma is a rare and very aggressive neoplasm that arises from the biliary epithelium, constitutes approximately 2% of all reported cancer, and accounts for about 3% of all gastrointestinal malignancies. Up to date, there are many modalities to diagnosis and treat with a range of sensitivity and specificity, and also the advantage and disadvantage of its modality. Cholangiocarcinoma has a poor prognosis. Surgical resection offers the only curative option and usually requires a major hepatic resection in addition to resection of the cholangiocarcinoma. Unfortunately, curative resection is possible in only about 30% of patients due to locally advanced disease, distant metastases or comorbidity in elderly patients. Even after resection, the recurrence rate is approximately 60%, resulting in a low 5-year overall survival (OS).

Patients with intra-hepatic Cholangiocarcinoma (ICC) have a very limited benefit from systemic chemotherapy, indeed, in unresectable cholangiocarcinoma Overall Survival with systemic chemotherapy is less than 1 year. Since most cholangiocarcinoma patients develop distant metastases at late stages only, locoregional therapy is an interesting therapeutic strategy.

Locoregional therapy studies in patients with intrahepatic cholangiocarcinoma employing radiofrequency ablation (RFA), transarterial chemoembolization (TACE) or external as well as internal radiation therapy yielded promising results in the last couple of years.

TACE is safe and may be effective for prolonging the survival of patients with nonresectable combined hepatocellular carcinoma (HCC) -cholangiocarcinoma, as compared with the historically reported survivals of these patients. Tumor vascularity is highly associated with tumor response. The patient survival period after TACE for combined HCC-cholangiocarcinoma is significantly dependent on tumor size, tumor vascularity, Child-Pugh class, and presence or absence of portal vein invasion.

Currently, few centers perform TACE therapy for unresectable Cholangiocarcinoma. Several European studies have reported the efficacy and safety TACE for ICC.

The establishment of a registry to obtain the majority of Cholangiocarcinoma cases treated with locoregional approach within and outside Europe can help the investigators evaluate a larger and non-ambiguous sample population. This would help the investigators evaluate the technical success rates, clinical success rates, feasibility and safety of TACE for ICC.

DETAILED DESCRIPTION:
Study Design: Prospective observational study

Primary objective: This is a data collection study where the main purpose is to collect information about the treatments that patients receive for their unresectable cholangiocarcinoma.

Secondary objectives: To create an international Registry including patients undergoing locoregional treatments, to correlate tumour characteristics with outcome, survival and prognosis; to identify criteria for guiding therapy including TACE, chemoinfusion and other locoregional treatments

Treatment modalities for TACE

Day -1 Doxorubicina 50-75 mg/mq has been charged onto 2 ml of 70-150 µm M1 microspheres at Pharmacy.

Day -1 : prehydration, antibiotic prophylaxis and setting up of a therapeutic scheme appropriate for analgesic prophylaxis (3-day duration) as previously reported 1 vial of tropisetron (diluted in 100ml of physiological solution) administered by slow drip Day 0: Upon admittance to the radiology room, the patient receive morphine hydrochloride 10 mgr diluted in 100 ml of salin solution i.v. (to be repeated one hour after the procedure and if necessary also after 6 hours).

Tropisetron i.v. if needed. Intra-arterial premedication with 2.5 mgr of verapamil 2.5 mgr diluted in 4 ml of normal saline solution followed by 4 ml of lidocaine 2%.

Selected arterial Infusion (considering tumor uptake and dominant disease) of doxorubicina 50-75 mg preloaded into 2 ml of 70-150 µm M1 microspheres.

Second infusion of doxorubicin at the same dose into 2 ml of 70-150 µm M1 microspheres can be administered in a further TACE (oncologist's planning of cure).

Day +30: The above procedure is repeated. Day +90: In case of response, a third administration following the above procedures will be repeated

Evaluation of response

Response must be assessed by repeating the following examinations at Day 30, Day 90 and Day 120 after start of treatment:

Chest-abdomen CAT scan with and without contrast medium (refer to Section 4). Evaluation will be based on the Response Evaluation Criteria In Solid Tumors (RECIST) cancer markers (CEA), Cancer Antigen (CA) 19.9)

Assessment of quality of life The Edmonton Symptom Assessment System (ESAS) is used to monitor health conditions and quality of life.

The questionnaire must be filled in by the patient unaided by family members or by health care personnel, over a period of about 15 minutes. Assessment of quality of life will be performed during the baseline visit and at Day 30, Day 60 and Day 120 from start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of cholangiocarcinoma will be established preoperatively by at least one of the following criteria: a) positive brush cytology or biopsy result obtained at the time of cholangiography; b) Fluorescence in situ hybridization demonstrating aneuploidy; c) serum CA 19-9 value greater than 100 U/mL in the presence of a radiographically characteristic malignant stricture in the absence of cholangitis.
2. Tumor is above the cystic duct and is unresectable.
3. Patient is a suitable candidate for the study by a radiation oncologist, a medical oncologist, and the liver surgeon
4. Maximum Eastern Cooperative Oncology Group performance status of 2 and a minimum daily caloric intake of 1200kcal.
5. No evidence of metastatic disease.
6. Between ages 18 - 75.
7. Patient must provide written informed consent.

Exclusion Criteria:

1. Patients with intrahepatic metastasis presenting liver involvement more than 75%
2. Patients with uncontrolled infections (sepsis)
3. Evidence of extrahepatic disease, including local lymph node metastasis (except peri-hilar nodes).
4. History of another malignancy diagnosed within 5 years, excluding "in situ" skin and cervical cancers, without metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-07; Primary Completion 2019-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
tumor response | 12 months
  CT scan evaluated with RECIST 1.1
overall survival | 12 months
  survival from start of treatment

SECONDARY OUTCOMES:
number adverse events | 4 months
  number of adverse events observed for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Giammaria Fiorentini, MD, Principal Investigator — International Group of Endovascular Oncology
Locations (1):
- Azienda Ospedaliera Ospedali Riuniti Marche Nord, Presidio Ospedaliero San Salvatore, Pesaro, Italy

REFERENCES:
- [Result] Aliberti C, Benea G, Tilli M, Fiorentini G. Chemoembolization (TACE) of unresectable intrahepatic cholangiocarcinoma with slow-release doxorubicin-eluting beads: preliminary results. Cardiovasc Intervent Radiol. 2008 Sep-Oct;31(5):883-8. doi: 10.1007/s00270-008-9336-2. Epub 2008 May 14. PMID 18478290
- [Result] Cantore M, Fiorentini G, Mambrini A, Rabbi C, Zamagni D, Carlone N, Manni A, Caudana R, Torri T. Regional combined with systemic chemotherapy in unresectable biliary tract cancers: a phase II study. J Exp Clin Cancer Res. 2003 Dec;22(4 Suppl):59-64. PMID 16767908
- [Derived] Fiorentini G, Mambrini A, Sarti D, Cantore M, Mulazzani L, Mattioli GM, Guadagni S. Hepatic intra-arterial and systemic chemotherapy followed by maintenance therapy for the treatment of cholangiocarcinoma. Hepat Oncol. 2017 Apr;4(2):45-53. doi: 10.2217/hep-2017-0001. Epub 2017 Aug 31. PMID 30191053
- See also: International group of endovascular oncology (IGEVO) website — http://igevo.jimdo.com/